CLINICAL TRIAL: NCT05946356
Title: The Relationship Between Psychological Wellbeing, Physical Activity, and Disability in Patients With Fibromyalgia: A Cross-Sectional Study
Brief Title: Psychological Wellbeing, Physical Activity, and Disability in Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: FIBRO8002023
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fibromyalgia patients: Participants will complete self-reported questionnaires to assess psychological wellbeing, physical activity, and disability.
  Interventions: Other: no intervention - cross-sectional observational only

INTERVENTIONS:
Other: no intervention - cross-sectional observational only — no intervention - cross-sectional observational only

SUMMARY:
This study aims to investigate the association between psychological wellbeing, physical activity, and disability in patients with fibromyalgia. Participants will complete self-reported questionnaires to assess psychological wellbeing, physical activity, and disability. The study will use descriptive statistics, correlation analysis, and multiple regression analysis to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* Age between 18 and 70 years old

Exclusion Criteria:

* Unable to complete self-reported questionnaires
* Presence of other chronic pain conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2023-11-25 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety, and Stress Scale (DASS) | Baseline
  epression, Anxiety, and Stress Scale (DASS) is a self-report questionnaire that is used to assess the severity of depression, anxiety, and stress. The DASS consists of 42 items that are scored on a scale of 0 to 3, with 0 indicating "not at all" and 3 indicating "severely." The total score for the DASS is the sum of the scores for the 42 items. A higher score indicates more severe symptoms of depression, anxiety, or stress.
International Physical Activity Questionnaire (IPAQ) | Baseline
  International Physical Activity Questionnaire (IPAQ) is a self-report questionnaire that is used to assess physical activity levels. The IPAQ consists of 7 questions that ask about the frequency, duration, and intensity of physical activity. The IPAQ can be used to assess physical activity levels in people of all ages and activity levels.
Fibromyalgia Impact Questionnaire (FIQ) | Baseline
  is a self-report questionnaire that is used to measure disability in patients with fibromyalgia. The FIQ consists of 21 items that ask about the impact of fibromyalgia on physical function, social function, and role function. The FIQ can be used to assess the severity of fibromyalgia and to monitor the effectiveness of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No